CLINICAL TRIAL: NCT07059221
Title: A Multicenter, Open-label Phase Ib/II Clinical Trial of SHR-A2102 Injection in Combination With Adebrelimab Injection, With or Without Other Anti-tumor Therapies, in Subjects With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Trial of SHR-A2102 With Adebrelimab With or Without Other Anti-tumor Therapies in Recurrent/MetastaticHead and Neck Squamous Cell Carcinoma Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-211
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A2102+Adebrelimab (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Adebrelimab
- SHR-A2102+Adebrelimab+Cetuximab (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Adebrelimab; Drug: Cetuximab

INTERVENTIONS:
Drug: SHR-A2102 — Administration by intravenous infusion
Drug: Adebrelimab — Administration by intravenous infusion
Drug: Cetuximab — Administration by intravenous infusion
  Arms: SHR-A2102+Adebrelimab+Cetuximab

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 with Adebrelimab with or without other Antitumor Therapy in Subjects with Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma.

To explore the reasonable dosage of SHR-A2102 for n Subjects with Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements.
2. The age of signing the informed consent is >= 18 years, regardless of gender.
3. Subject with advanced or distant metastatic squamous cell carcinoma of the head and neck confirmed by histology or cytology.
4. Tumors with primary foci located in the oropharynx, oral cavity, hypopharynx and larynx.
5. Provide archived or fresh tumor tissue for test.
6. At least one measurable lesion according to RECIST v1.1 criteria.
7. The ECOG score is 0 or 1.
8. Expected survival ≥12 weeks.
9. Good level of organ function.
10. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods.

Exclusion Criteria:

-

1. Subjects will not be screened if they meet any of the following conditions:

1. Primary tumor located in the nasopharynx, salivary glands, sinuses, skin, or squamous cell carcinoma of unknown primary origin;
2. Locally advanced patients who are candidates for curative surgery or local therapy and have the intention to undergo such treatment;
3. Presence of necrotic lesions or significant tumor invasion into adjacent organs or blood vessels, as assessed by the investigator, posing a high risk of major bleeding.

2. Known hypersensitivity to the investigational drug or any of its excipients, or a history of severe allergic reactions to other monoclonal antibodies.

3. Prior treatments or medications before the first dose of the study drug:

1. Use of any investigational drug within 4 weeks before the first dose;
2. Concurrent enrollment in another clinical trial, unless it is an observational (non-interventional) study or follow-up in an interventional study;
3. Last dose of anticancer therapy (including chemotherapy, biologic therapy, immunotherapy, targeted therapy, etc.) within 4 weeksbefore the first dose; for small-molecule targeted drugs, within 2 weeks or 5 half-lives (whichever is longer); traditional Chinese medicine with antitumor indications within 2 weeks before the first dose.

4. Active autoimmune disease or a history of autoimmune disorders. 5、 Residual toxicity from prior anticancer therapy not resolved to ≤Grade 1 (CTCAE v5.0) (except for non-safety risks, such as alopecia) or not meeting the inclusion/exclusion criteria.

6、 Uncontrolled or symptomatic active CNS metastases. 7、 Symptomatic visceral metastases with imminent life-threatening complications .

8、 Known or suspected interstitial lung disease (ILD) or severe pulmonary conditions.

9、 Other active malignancies within 3 years before study entry. 10、 Clinically significant cardiovascular disease. 11、 Active or chronic infections of clinical significance. 12、 Pregnancy or lactation. 13、 Other factors that, in the investigator's judgment, may lead to premature study discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
RP2D | through phase IB completion, an average of 5 years
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in Phase IB stages
Incidence and severity of AE(DLT) | from Day1 to 90 days after last dose
  According to NCI-CTCAE v5.0 evaluation criteria from Day 1 to 90 days after last dose
ORR | 5 years after the last subject was enrolled in the group
  efficacy was assessed every 6 weeks as determined by RECIST1.1

SECONDARY OUTCOMES:
DCR | 5 years after the last subject was enrolled in the group
  Since C1D1 every 6 weeks w and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
DOR | 5 years after the last subject was enrolled in the group
  Since C1D1 every 6 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
PFS(Investigator evaluation) | 5 years after the last subject was enrolled in the group
  Since C1D1 every 6 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
OS(Investigator evaluation) | 5 years after the last subject was enrolled in the group
  Since C1D1 and death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided